CLINICAL TRIAL: NCT02513290
Title: Quality of Life in Patients With Allergic Rhinitis: a Clinical Trial Comparing the Use of Bilastine Versus Loratadine
Brief Title: Quality of Life in Patients With Allergic Rhinitis: Clinical Trial With Bilastine or Loratadine
Acronym: QolRhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade do Sul de Santa Catarina (Other Government)
Responsible Party: Principal Investigator, Jane da Silva, PhD, Universidade do Sul de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTBixLo
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Allergic Rhinitis
Keywords: quality of life; allergic rhinitis; bilastine; loratadine; clinical trial
MeSH Terms: conditions — Rhinitis, Allergic | interventions — bilastine; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilastine group (Experimental): Bilastine 20 mg administered once a day for ten days.
  Interventions: Drug: Bilastine
- Loratadine group (Experimental): Loratadine 10 mg administered once a day for ten days.
  Interventions: Drug: Loratadine

INTERVENTIONS:
Drug: Bilastine
  Other Names: Alektos
  Arms: Bilastine group
Drug: Loratadine
  Other Names: Claritin; Histadin; Loranil; Loritil; Loralerg
  Arms: Loratadine group

SUMMARY:
The purpose of this study was to verify whether there were differences in health-related quality of life of patients with allergic rhinitis treated with bilastine 20 mg compared to those treated with loratadine 10 mg.

DETAILED DESCRIPTION:
This was a prospective randomized double-blinded study, in which patients were recruited from august 2013 until august 2014. Outpatients attended in 4 otolaryngology clinics from Criciúma, state of Santa Catarina, Brazil were invited to participate of the study. They were aged between 18 and 63 years. Seventy-three patient were included, of whom 36 were treated with loratadine 10 mg and 37 with bilastine 20 mg with medication administered once a day for ten days. The primary outcome was quality of life, assessed by the modified Rhinoconjunctivitis Quality of Life Questionnaire (RQLQm), which was applied at baseline and after 10 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of allergic rhinitis (a typical history of rhinitis symptoms: coryza, sneezing, nasal obstruction, nasal itching, and eye symptoms, and hypersensitivity tests for specific IgE measured by Radioallergosorbent Test (RAST) or skin tests
* patients classified as with intermittent rhinitis (symptoms during less than 4 days per week) or persistent rhinitis (symptoms during more than 4 days per week) of moderate to severe intensity (annoyance impairing the quality and quantity of sleep and interfering with daily activities)

Exclusion Criteria:

* pregnancy or breast-feeding;
* non-allergic rhinitis (vasomotor, infectious or drug-induced);
* known hypersensitivity to antihistamines;
* clinical disorders that might affect the assessment;
* nasal diseases that could lead to complete blockage or one of the nostrils blockage, such as tumors or septal deviation;
* therapy with immunotherapy;
* use of antihistamines or disodium cromoglycate within the past four weeks;
* use of topical or systemic corticosteroids, immunosuppressants or any investigational drug within the last two weeks;
* use of topical antihistamines or nasal decongestants within the last 48 hours;
* use of deposit steroid within the last month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Quality of life in patients with allergic rhinitis | 10 days
  Application of the modified Rhinoconjunctivitis Quality of Life Questionnaire (RQLQm)

CONTACTS AND LOCATIONS:
Overall Officials: Jane da Silva, PhD, Principal Investigator — Universidade do Sul de Santa Catarina

REFERENCES:
- [Background] Juniper EF, Thompson AK, Ferrie PJ, Roberts JN. Validation of the standardized version of the Rhinoconjunctivitis Quality of Life Questionnaire. J Allergy Clin Immunol. 1999 Aug;104(2 Pt 1):364-9. doi: 10.1016/s0091-6749(99)70380-5. PMID 10452758
- [Background] Carter NJ. Bilastine: in allergic rhinitis and urticaria. Drugs. 2012 Jun 18;72(9):1257-69. doi: 10.2165/11209310-000000000-00000. PMID 22686617
- [Background] Nascimento Silva M, Naspitz C, Sole D. Evaluation of quality of life in children and teenagers with allergic rhinitis: adaptation and validation of the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ). Allergol Immunopathol (Madr). 2001 Jul-Aug;29(4):111-8. doi: 10.1016/s0301-0546(01)79042-8. PMID 11674923
- [Background] Bachert C, Kuna P, Sanquer F, Ivan P, Dimitrov V, Gorina MM, van de Heyning P, Loureiro A; Bilastine International Working Group. Comparison of the efficacy and safety of bilastine 20 mg vs desloratadine 5 mg in seasonal allergic rhinitis patients. Allergy. 2009 Jan;64(1):158-65. doi: 10.1111/j.1398-9995.2008.01813.x. PMID 19132976
- [Background] Van Cauwenberge P, Juniper EF. Comparison of the efficacy, safety and quality of life provided by fexofenadine hydrochloride 120 mg, loratadine 10 mg and placebo administered once daily for the treatment of seasonal allergic rhinitis. Clin Exp Allergy. 2000 Jun;30(6):891-9. doi: 10.1046/j.1365-2222.2000.00914.x. PMID 10848909